CLINICAL TRIAL: NCT04860310
Title: Panoramic Presentation and Tolerance Mechanism of Human Endometrium Based on Tiangui Theory
Status: Completed | Type: Observational
Sponsor: Heilongjiang University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Xiaoke Wu, Director of Obstetrics and Gynecology Department, Heilongjiang University of Chinese Medicine
Other Study IDs: MOM
Record Dates: First submitted 2021-04-06; First posted 2021-04-26 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Endometrium; Senility

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- 21 years old group
  Interventions: Procedure: Endometrial biopsy
- 28 years old group
  Interventions: Procedure: Endometrial biopsy
- 35 years old group
  Interventions: Procedure: Endometrial biopsy
- 42 years old group
  Interventions: Procedure: Endometrial biopsy
- 49 years old group
  Interventions: Procedure: Endometrial biopsy

INTERVENTIONS:
Procedure: Endometrial biopsy — Subjects need to collect 5ml whole blood (EDTA or heparin anticoagulant) once in the morning on an empty stomach. Endometrial tissue samples were taken during a complete 28-day menstrual cycle, a total of 6 times, and blood was taken to measure the level of gonadal hormones before each sampling.

SUMMARY:
Detailed Description:In the process of women's menstrual cycle, there are different physiology at different time points in a cycle.

Change, investigators select women with a menstrual cycle of 28 days and take samples every 3 days.

Day 4, Day 7, Day 10, Day 13, Day 16, Day 19, Day 22, Day 25, Day 28 days, a total of 10 time points, 20 healthy women were selected, and the transcription, Protein and phosphorylation proteomics, systematically integrated analysis; at the same time, 20 subjects were classified by age group Divide into 4 groups, 21-year-old group, 28-year-old group, 35-year-old group, and 42-year-old group. At the same time, investigators then analyze the differences in the receptivity of the endometrium of different ages.

The experimental design groups are: 21-year-old group, 28-year-old group, 35-year-old group, 42-year-old group, Each group includes D1 group Vs D4 group Vs D7 group Vs D10 group Vs D13 group Vs D16 group Vs D19 group Vs D22 group Vs D25 group Vs D28 group; in phosphorylation modification omics, different time points are compared with each other, Look for transcripts, proteins and phosphorylated proteins that change significantly during the cycle of change. Analyze phosphorylation modification An important role for changing proteins and an important role for cycle changes.

The experiment quantified the proteome and protein acylation modification through TMT (Tandem Mass Tag), and passed GO, KEGG Pathway, Localization, Functional enrichment analysis, Cluster analysis Bioinformatics analysis

ELIGIBILITY:
Inclusion criteria:

1. The subject's infertility factors are only male factors and/or fallopian tube factors;
2. Age: 21/28/35/42/49 years old (calculated according to the birthday month of the Gregorian calendar, no more than 6 months before and after);
3. Body mass index (weight/height square)=23～25kg/m2;
4. The menstrual cycle is 28+/-1 days (that is, the menstruation is 2-3 days in advance of each month), and the consistency of the past 6 consecutive months (not more than 1 day before and after, that is, 27-29 days);
5. Women with a history of pregnancy are preferred;
6. Asexual life during the study period;
7. No IUD is placed in the uterine cavity;
8. Volunteer to participate in the experiment and sign the informed consent form.

Exclusion criteria:

1. Women who have a history of miscarriage;
2. Women during pregnancy and breastfeeding;
3. Mentally ill;
4. Those who have had oral contraceptives or hormonal drugs in the past three months;
5. Combined with serious primary diseases such as cardiovascular, cerebrovascular, liver, kidney and hematopoietic system;
6. Subjects who have participated in other drug clinical trials within six months;
7. Those who have poor compliance and the investigator thinks it is inappropriate to participate in this clinical trial.

Ages: 21 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The subject is a healthy woman aged 21/28/35/42/49 years old, BMI=23～25kg/m2, and her menstrual cycle is 28+/-1 day (that is, 2-3 days in advance of each month) , And consistent for the past 6 consecutive months (no more than 1 day before and after, that is, 27-29 days), no IUD was placed in the uterine cavity.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2020-07-08 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2021-09-05 (Actual)

PRIMARY OUTCOMES:
Panorama of the endometrium | Menstrual cramps 24 hours, the seventh day of menstruation, LH peak, 72 hours after the peak, the 21st day of menstruation, the 28th day of menstruation
  Discovery of inner membrane receptive proteins and pathways

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology,First Affliated Hospital,Heilongjiang University of Chinese Medicine ., Harbin, Heilongjiang, China